CLINICAL TRIAL: NCT00005291
Title: Clinical Epidemiology of Asthma in An HMO
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 2013; R29HL041039 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-06

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To provide information on morbidity and health care utilization for asthma for a large, well-defined population over a 20 year period.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is the second most common chronic respiratory disorder seen by physicians in outpatients, and in 1988 was estimated to be the primary or secondary cause of 9.3 percent of all physician office visits for ambulatory medical care in the United States. Reports citing increased asthma morbidity and mortality in this country and abroad have intensified interest in this disorder. Investigations into possible explanations for these increases, however, have been hampered by the lack of good longitudinal data on the incidence, prevalence, and health care utilization associated with asthma, and by the lack of generally accepted diagnostic criteria for defining the disease.

DESIGN NARRATIVE:

Use of the Kaiser-Permanente Northwest Region data base allowed an examination of the secular trends in the prevalence and incidence of physician-diagnosed asthma and asthma-like disorders in inpatient and outpatient populations over a 20 year period, health care utilization and temporal changes in utilization patterns for asthma, and the natural history of asthma in selected subpopulations. Demographic factors examined were limited to age and sex.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1988-07; Study Completion 2003-04 (Actual)

REFERENCES:
- [Background] Vollmer WM, Buist AS, Osborne ML. Twenty year trends in hospital discharges for asthma among members of a health maintenance organization. J Clin Epidemiol. 1992 Sep;45(9):999-1006. doi: 10.1016/0895-4356(92)90115-4. PMID 1432028
- [Background] Osborne ML, Vollmer WM, Buist AS. Diagnostic accuracy of asthma within a health maintenance organization. J Clin Epidemiol. 1992 Apr;45(4):403-11. doi: 10.1016/0895-4356(92)90041-k. PMID 1569436
- [Background] Osborne ML, Vollmer WM, Johnson RE, Buist AS. Use of an automated prescription database to identify individuals with asthma. J Clin Epidemiol. 1995 Nov;48(11):1393-7. doi: 10.1016/0895-4356(95)00065-8. PMID 7490602
- [Background] Vollmer WM, Osborne ML, Buist AS. Temporal trends in hospital-based episodes of asthma care in a health maintenance organization. Am Rev Respir Dis. 1993 Feb;147(2):347-53. doi: 10.1164/ajrccm/147.2.347. PMID 8430957
- [Background] Vollmer WM, Osborne ML, Buist AS. 20-year trends in the prevalence of asthma and chronic airflow obstruction in an HMO. Am J Respir Crit Care Med. 1998 Apr;157(4 Pt 1):1079-84. doi: 10.1164/ajrccm.157.4.9704140. PMID 9563722
- [Background] Osborne ML, Vollmer WM, Buist AS. Periodicity of asthma, emphysema, and chronic bronchitis in a northwest health maintenance organization. Chest. 1996 Dec;110(6):1458-62. doi: 10.1378/chest.110.6.1458. PMID 8989061